CLINICAL TRIAL: NCT03305445
Title: A Multi-center Phase Ib/II Trial of Nivolumab/Ipilimumab-Primed Immunotransplant for Relapsed/Refractory Diffuse Large B Cell Lymphoma Patients.
Brief Title: Nivolumab/Ipilimumab-Primed Immunotransplant for DLBCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Joshua Brody, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-2164
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: Immunotransplant; Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Nivolumab; Ipilimumab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: This multi-center study open-label trial will enroll a single cohort of relapsed/refractory diffuse large B cell lymphoma (DLBCL) patients whom are ineligible for autologous stem cell transplant (ASCT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pts with Diffuse Large B Cell Lymphoma (Experimental): Patients with DLBCL not eligible for autologous stem cell transplant. All patients will receive dual checkpoint blocking antibody (DCBA) therapy of ipilimumab and nivolumab given at three week intervals, two times before, and two times following "immunotransplant" in which T cells (in whole PBMCs) are cryopreserved and re-infused (adoptive T cell transfer or ATCT) following lymphodepleting chemotherapy regimen, currently being employed in adoptive T cell therapies.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab (1mg/kg)
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab (3mg/kg)
  Other Names: Opdivo

SUMMARY:
This multi-center study open-label trial will enroll a single cohort of relapsed/refractory diffuse large B cell lymphoma (DLBCL) patients whom are ineligible for autologous stem cell transplant (ASCT) due to 1) insensitivity to salvage chemotherapy, or 2) inability to tolerate high-dose myeloablative chemotherapy. All patients will receive dual checkpoint blocking antibody (DCBA) therapy with established doses currently being used in phase III trials of ipilimumab (1mg/kg) and nivolumab (3mg/kg) given at three week intervals, two times before, and two times following "immunotransplant" in which T cells (in whole PBMCs) are cryopreserved and re-infused (adoptive T cell transfer or ATCT) following lymphodepleting chemotherapy regimen, currently being employed in adoptive T cell therapies.

DETAILED DESCRIPTION:
First 6 patients will be part of Phase Ib. Phase Ib and Phase II: Will occur sequentially. Phase II will proceed only if toxicity is acceptable as determined in Phase Ib.

ELIGIBILITY:
Inclusion Criteria:

1. Have pathologically confirmed DLBCL on biopsy.
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be ≥18 years of age on day of signing informed consent
4. Have a performance status of 0 or 1 on the ECOG Performance Scale
5. Demonstrate adequate organ function at time of screening as defined in Table 2 below, all screening labs should be performed within 14 days of treatment initiation.

   Table 2 Adequate Organ Function Laboratory Values System Laboratory Value Hematologica Absolute neutrophil count (ANC) ≥1,000 /mcL Platelets ≥25,000 / mcL Hemoglobin ≥8 g/dL Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤2.0 X upper limit of normal (ULN) OR

   ≥60 mL/min for subject with creatinine levels > 2.0 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR

   ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

   Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT is within therapeutic range of intended use of anticoagulants

   ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PTT is within therapeutic range of intended use of anticoagulants a Patients with cytopenias attributable to bone marrow lymphomatous bone marrow involvement per current bone marrow biopsy may be enrolled if other inclusion criteria are met.

   b Creatinine clearance should be calculated per institutional standard.
6. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of DCBA. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Female subjects of childbearing potential must be willing to use an adequate method of contraception. Contraception should be used for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
8. Male subjects of childbearing potential must agree to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.
9. Patients who did not achieve a PR or CR as per the Lugano criteria following at least 1 cycle of platinum-based salvage chemotherapy, or patients not eligible for platinum-based therapy or BEAM induction therapy due to decreased ejection fraction (<40%).
10. There is no upper age restriction.
11. Patients whom have undergone previous autologous stem cell transplant, and have recurrent or residual disease are eligible for this trial.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to ipilimumab or nivolumab or any of their excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 28 days prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 28 days earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or lymphomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 28 days prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include lymphomatous meningitis, which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a systemic treatment. Subjects on stable dose of corticosteroids less than or equivalent to 10mg of prednisone daily for more than 3 months may be enrolled, and continue their stable dose through treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment (roughly two and a half years after enrollment).
15. HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen.
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. History of allogeneic stem-cell (or other organ) transplantation.
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | 3 months
  DLTs recorded and graded according to NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. for Phase 1B part of study
Completion Remission (CR) Rate | 3 months
  The proportion of patients who have achieved complete remission as per Lugano criteria which is complete metabolic response even with a persistent mass.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  PFS will be estimated using the method of Kaplan-Meier where PFS is defined as the time from Adoptive T cell transfer (ATCT) until the first recurrence or progression of disease as per Lugano criteria (3), or date of death if the subject dies from any cause before progression is documented.
Overall Survival (OS) | 2 years
  OS from the time of ATCT (D0) until recorded date of death.
IgVH level | 2 years
  Rate and time to achieving molecular remission as determined by serum analysis for persistent IgVH by PCR
Delayed CR | 2 years
  Delayed CR defined as the proportion of patients who achieved CR reported as a percentage of the total number of subjects enrolled for both FA and PP populations.
Overall Response Rate (ORR) | 2 years
  ORR, defined as CR+PR+SD (complete remission + partial remission + stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Brody, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No